CLINICAL TRIAL: NCT00255580
Title: Placebo-Controlled, Double Blind Trial of Medicinal Cannabis in Painful HIV Neuropathy
Brief Title: Medicinal Cannabis for Painful HIV Neuropathy
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Center for Medicinal Cannabis Research (Other)
Responsible Party: Ronald J. Ellis, M.D., Ph.D., University of California, San Diego
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: C00-SD-104
Record Dates: First submitted 2005-11-17; First posted 2005-11-21 (Estimated); Last update posted 2008-02-28 (Estimated); Status verified 2008-02

CONDITIONS: Neuropathic Pain
Keywords: neuropathy; cannabis; marijuana; HIV; DSPN
MeSH Terms: conditions — Neuralgia; Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Active cannabis (1-8% THC by weight)
  Interventions: Drug: Smoked cannabis
- 2 (Placebo Comparator): Placebo cannabis
  Interventions: Drug: Smoked cannabis

INTERVENTIONS:
Drug: Smoked cannabis

SUMMARY:
The purpose of this study is to determine if medicinal cannabis (marijuana) is safe and effective for treating pain in individuals with HIV-associated distal, sensory-predominant polyneuropathy (DSPN).

DETAILED DESCRIPTION:
Peripheral neuropathy occurs in over 30% of patients with HIV infection, making it among the most common neurological complications of HIV infection. Nucleoside analogues such as ddI and d4T, key components of modern, potent, combination antiretroviral therapies (ART), are also neurotoxic and contribute to the frequent occurence of painful neuropathy. By using treatment with available non-narcotic analgesic and adjunctive pain medications, approximately half of patients with painful HIV neuropathy obtain sufficient pain control.

On the first day each study week (active or placebo), participants will follow a specific titration procedure to achieve the optimal dose. This optimal dose will then be continued for the duration of the treatment week. Participants will undergo a 2-week washout period, after which they crossover to the other arm (active or placebo) and will again repeat the dose titration and dose maintenance procedures.

Comparison: Active cannabis doses ranging from 2-8% THC will be compared to placebo for the reduction of neuropathic pain.

ELIGIBILITY:
Inclusion Criteria:

* Documented HIV infection
* Meets clinical and electrodiagnostic criteria for HIV-associated DSPN at entry
* Daily pain for at least three consecutive months with an average daily pain magnitude score of at least 5 on the Descriptor Differential Scale
* Inadequate pain relief with prior treatment for painful HIV neuropathy using drugs from at least two different classes of pain-modifying agents (NSAIDS, low-potency opioids, high-potency opioids, sodium channel blockers, other adjunctive pain treatments)
* Age 21-65 years
* Stable use of opioid and non-opioid analgesic medications during the two weeks prior to study entry

Exclusion Criteria:

* Positive urine toxicology screen for cannabinoids during the "wash-in" week prior to initiating study treatment
* Recent (i.e. during the month prior to study entry) history of marijuana use more than twice a week
* Previous psychosis with or intolerance to cannabinoids
* A lifetime history (ever) of dependence on cannabis
* Meeting criteria for alcohol or drug dependence within the last 12 months
* Active, major psychiatric disorder likely, in the investigator's opinion, to interfere with adherence to the study protocol
* Active AIDS-defining opportunistic disease (a history of AIDS-defining opportunistic disease which is no longer active or progressing will not be grounds for exclusion)
* Diabetes mellitus, renal failure with uremia, alcohol abuse, previous spinal surgery, or other documented causes of neuropathy or neuropathic pain
* Pulmonary disease of sufficient severity to require the use of supplemental oxygen
* Asthma
* Life expectancy less than 6 weeks or an active, acute illness likely to interfere with completion of the study protocol
* Pregnancy
* Failure to use adequate birth control in an individual with reproductive potential
* Minority status (less than 21 years), or persons over age 65 years

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2001-09; Primary Completion 2006-11 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Descriptor Differential Scale (DDS) | Baseline, Post-treatment

SECONDARY OUTCOMES:
Changes in the use of opioid and non-opioid analgesics | Post-Treatment
Changes in measures of everyday functioning and subject-perceived quality of life | Baseline, Post-Treatment
Adverse effects | Post-Treatment
Adverse cognitive effects as assessed by neuropsychological testing. | Baseline, Post-Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Ellis, M.D., Ph.D., Principal Investigator — University of California, San Diego
Locations (1):
- UC San Diego, Hillcrest Medical Center, San Diego, California, United States

REFERENCES:
- See also: Center for Medicinal Cannabis Research — http://cmcr.ucsd.edu
- See also: HIV Neurobehavioral Research Center — http://hnrc.ucsd.edu